CLINICAL TRIAL: NCT05672563
Title: Cesarean Scar Evaluation Using Saline Infusion Sonography in Women With Previous Pregnancy in Scar
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0298-22-ASF
Record Dates: First submitted 2023-01-01; First posted 2023-01-05 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2022-12

CONDITIONS: Uterus; Scar
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Intervention Model Description: Prospective cohort study in a tertiary referral center. Investigators evaluated the procedure on a group of 40 participants that are invited to our unit for evaluation of cesarean scar by using a saline-infused sonography examination. Secondly, the medical records of all identified cases are retrospectively reviewed and the CSPs are classified into three subgroups according to the level of CSP sac herniation proposed by the Delphi criteria.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- women with previous CSP (Experimental): experimental: women with previous cesarean scar pregnancy that are invited to our unit for sonographic evaluation.
  Interventions: Drug: Saline infusion sonography for evaluation of cesarean scar

INTERVENTIONS:
Drug: Saline infusion sonography for evaluation of cesarean scar — The intervention included the usage of balloon-less GIS catheter with a soft tapered tip inserted into the endocervical canal, with no use of a tenaculum or a cervical dilatator. Normal saline is slowly introduced into the uterine cavity via the catheter until achieving satisfactory distension and visualization of the uterine cavity using trans-vaginal ultra-sonographic imaging.
  Other Names: Saline infusion

SUMMARY:
Evaluation of cesarean scar using saline-infused sonography in women with history of cesarean scar pregnancy.

DETAILED DESCRIPTION:
Over the past few decades, cesarean delivery rates worldwide have risen considerably. The surgery may lead to deficient uterine scar healing, thinning of the myometrium and formation of cesarean scar defects or uterine scar niche. The prevalence of clinically relevant cesarean scar defects is unclear and has been reported between 20-88%, it is identified by using transvaginal ultrasound or saline-infused sonography in non-pregnant patients. Women may be asymptomatic or present a wide gynecologic sequela including cesarean scar pregnancy, abnormal uterine bleeding, dysmenorrhea, chronic pelvic pain, infertility, and increased risk of complications during gynecologic procedures such as uterine evacuation and insertion of intrauterine device.

Cesarean scar pregnancy (CSP) is defined as an early pregnancy implantation in the scar from a prior cesarean delivery. This pregnancy is implanted in a fibrous scar tissue and may lead to substantial risk for severe maternal morbidity such as adherent placenta, second or third trimester uterine dehiscence or rupture, severe maternal bleeding, and adherence to adjacent tissues. The prevalence of scar pregnancy is reported to be between 1:1800-2500 pregnancies, with increasing diagnosis in the last decade due to increasing use of transvaginal ultrasound early in pregnancy and possible increased physician awareness of this condition.

The ultrasound criteria for CSP have been redefined recently, and now propose transvaginal ultrasound as the imaging technique of choice at this early stage. In 2022, the Niche Task-force convened a Delphi consensus to develop a standardized sonographic evaluation and reporting system for a CSP in the first trimester. According to this consensus, CSPs were classified into three subgroups, Subgroup A in which the largest part of the gestational sac protruded towards the uterine cavity, subgroup B in which the largest part of the gestational sac was embedded in the myometrium, and subgroup C in which the gestational was partially located outside the outer contour of the cervix or uterus. This sonographic classification has yet to be validated clinically.

In the present report the investigators aim to evaluate the uterine cavity and potential cesarean scar defects or niche in women with history of CSP using saline infused sonography. In the second stage of the research, we will classify the past cesarean pregnancies according to the new Delphi criteria and examine correlation between the different CSP subgroups and presence of cesarean scar defects.

ELIGIBILITY:
Inclusion Criteria:

* women with history of cesarean scar pregnancy

Exclusion Criteria:

* ongoing pregnancy
* vaginal bleeding
* active or suspected inflammation of genital tract including pelvic inflammatory disease
* women engaged in unprotected intercourse
* presence of intra-uterine device contraception

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Uterine niche | through study completion, an average of 6 months
  Number of participants who underwent saline infused sonography and have evidence of cesarean scar defects/ uterine niche.

CONTACTS AND LOCATIONS:
Overall Officials: Yaakov Melcer, Professor, Principal Investigator — Assaf-Harofeh Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Betran AP, Ye J, Moller AB, Zhang J, Gulmezoglu AM, Torloni MR. The Increasing Trend in Caesarean Section Rates: Global, Regional and National Estimates: 1990-2014. PLoS One. 2016 Feb 5;11(2):e0148343. doi: 10.1371/journal.pone.0148343. eCollection 2016. PMID 26849801
- [Background] Jordans IPM, de Leeuw RA, Stegwee SI, Amso NN, Barri-Soldevila PN, van den Bosch T, Bourne T, Brolmann HAM, Donnez O, Dueholm M, Hehenkamp WJK, Jastrow N, Jurkovic D, Mashiach R, Naji O, Streuli I, Timmerman D, van der Voet LF, Huirne JAF. Sonographic examination of uterine niche in non-pregnant women: a modified Delphi procedure. Ultrasound Obstet Gynecol. 2019 Jan;53(1):107-115. doi: 10.1002/uog.19049. PMID 29536581
- [Background] Feldman N, Maymon R, Jauniaux E, Manoach D, Mor M, Marczak E, Melcer Y. Prospective Evaluation of the Ultrasound Signs Proposed for the Description of Uterine Niche in Nonpregnant Women. J Ultrasound Med. 2022 Apr;41(4):917-923. doi: 10.1002/jum.15776. Epub 2021 Jul 1. PMID 34196967
- [Background] Tower AM, Frishman GN. Cesarean scar defects: an underrecognized cause of abnormal uterine bleeding and other gynecologic complications. J Minim Invasive Gynecol. 2013 Sep-Oct;20(5):562-72. doi: 10.1016/j.jmig.2013.03.008. Epub 2013 May 14. PMID 23680518
- [Background] Society for Maternal-Fetal Medicine (SMFM). Electronic address: pubs@smfm.org; Miller R, Timor-Tritsch IE, Gyamfi-Bannerman C. Society for Maternal-Fetal Medicine (SMFM) Consult Series #49: Cesarean scar pregnancy. Am J Obstet Gynecol. 2020 May;222(5):B2-B14. doi: 10.1016/j.ajog.2020.01.030. Epub 2020 Jan 21. PMID 31972162
- [Background] Timor-Tritsch IE, Monteagudo A, Cali G, D'Antonio F, Kaelin Agten A. Cesarean Scar Pregnancy: Diagnosis and Pathogenesis. Obstet Gynecol Clin North Am. 2019 Dec;46(4):797-811. doi: 10.1016/j.ogc.2019.07.009. PMID 31677755
- [Background] Timor-Tritsch IE, Monteagudo A, Cali G, Palacios-Jaraquemada JM, Maymon R, Arslan AA, Patil N, Popiolek D, Mittal KR. Cesarean scar pregnancy and early placenta accreta share common histology. Ultrasound Obstet Gynecol. 2014 Apr;43(4):383-95. doi: 10.1002/uog.13282. PMID 24357257
- [Background] Timor-Tritsch IE, Horwitz G, D'Antonio F, Monteagudo A, Bornstein E, Chervenak J, Messina L, Morlando M, Cali G. Recurrent Cesarean scar pregnancy: case series and literature review. Ultrasound Obstet Gynecol. 2021 Jul;58(1):121-126. doi: 10.1002/uog.23577. PMID 33411387
- [Background] Cali G, Timor-Tritsch IE, Forlani F, Palacios-Jaraquemada J, Monteagudo A, Kaelin Agten A, Flacco ME, Khalil A, Buca D, Manzoli L, Liberati M, D'Antonio F. Value of first-trimester ultrasound in prediction of third-trimester sonographic stage of placenta accreta spectrum disorder and surgical outcome. Ultrasound Obstet Gynecol. 2020 Apr;55(4):450-459. doi: 10.1002/uog.21939. PMID 31788885
- [Background] Jordans IPM, Verberkt C, De Leeuw RA, Bilardo CM, Van Den Bosch T, Bourne T, Brolmann HAM, Dueholm M, Hehenkamp WJK, Jastrow N, Jurkovic D, Kaelin Agten A, Mashiach R, Naji O, Pajkrt E, Timmerman D, Vikhareva O, Van Der Voet LF, Huirne JAF. Definition and sonographic reporting system for Cesarean scar pregnancy in early gestation: modified Delphi method. Ultrasound Obstet Gynecol. 2022 Apr;59(4):437-449. doi: 10.1002/uog.24815. PMID 34779085